CLINICAL TRIAL: NCT02185456
Title: Validation of a Novel Diagnostic, Prognostic Assay for Bacterial Vaginosis
Acronym: BV-LbRC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Robert A. Akins, Principal investigator-coinvestigator, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: R21AI111103-01 (NIH); R21AI111103-01 (NIH)
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Metronidazole; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Healthy (No Intervention): Patients with no history of bacterial vaginosis. These women will be monitored monthly and with daily self swabs.
- G1 BV in clinical & molecular remission (Active Comparator): Patients will receive standard of care intervention, oral metronidazole 500 mg twice a day for 7 days. They will then be monitored to confirm that initial BV treatment was effective by Nugent and Amsel, and by the qPCR test (LbRC). These will be monitored with monthly visits and daily self swabs. Those who recur with symptomatic BV may enroll in the B2 arm for more aggressive treatment.
  Interventions: Drug: Standard of care
- G2. Molecular conversion subarm (Experimental): Half of G1 patients who convert to poor qPCR test results while remaining asymptomatic will be randomized into this G2 arm and receive intervention: 750 mg metronidazole/ 200 mg miconazole vaginal suppository daily for 7 days, with continued monthly visits and daily swabs.
  Interventions: Drug: 750 mg metronidazole/ 200 mg miconazole vaginal suppository; Drug: Standard of care
- B1 Initially poor qPCR responders (Active Comparator): The B1 arm are patients who enter remission after standard of care treatment, oral metronidazole 500 mg twice a day for 7 days, but who have poor initial qPCR scores. Half of such patients will be randomized into B1, half into B2. B1 patients will be monitored with monthly visits and via daily swabs, but will receive no further treatment while BV negative. Patients who recur with BV may enroll as B2 patients for more aggressive treatment.
  Interventions: Drug: Standard of care
- B2 BV Remission to conversion (Experimental): A subgroup of B1 patients who convert to consistently poor qPCR scores during the study (conversion) will be randomized into Arm B2 and receive intervention: 750 mg metronidazole/ 200 mg miconazole vaginal suppository daily for 7 days. These patients will continue monthly visits and daily self swabs. B2 patients who recur with symptomatic BV will be dropped from the study and given other options for therapy.
  Interventions: Drug: 750 mg metronidazole/ 200 mg miconazole vaginal suppository; Drug: Standard of care

INTERVENTIONS:
Drug: 750 mg metronidazole/ 200 mg miconazole vaginal suppository — The higher dose 750 mg metronidazole/ 200 mg miconazole vaginal suppository will be given to patients who were refractory to the standard of care therapy, oral metronidazole 500 mg twice a day for 7 days, and to asymptomatic patients in a randomized arm, who show poor responses based on the qPCR test result.
  Arms: B2 BV Remission to conversion; G2. Molecular conversion subarm
Drug: Standard of care — oral metronidazole 500 mg twice a day for 7 days
  Other Names: Flagyl
  Arms: B1 Initially poor qPCR responders; B2 BV Remission to conversion; G1 BV in clinical & molecular remission; G2. Molecular conversion subarm

SUMMARY:
Bacterial vaginosis (BV) is the commonest form of vaginitis worldwide, affecting millions of women. Unfortunately, recurrence rates of symptomatic BV remain extremely high, 30% at three months and 70-80% within a year. Given the paucity of information and data regarding pathogenesis of BV, the etiopathogenesis of recurrent bacterial vaginosis remains unknown. Accordingly, reliable, proven treatment regimens for Recurrent Bacterial Vaginosis (RBV) are not available.

In 2013, the investigators published two manuscripts documenting a new qPCR based approach to BV diagnosis and potentially prognosis. The method (LbRC) measures the content of lactobacilli in vaginal samples, relative to total bacterial load. The first goal of this study are to validate that this metric is a reliable diagnostic of BV, by determining sensitivities and specificities relative to Nugent scores and Amsel criteria of healthy women and BV patients. A high LbRC score (3-4) corresponds to a healthy state. The second goal is to determine whether empirically determined "low" LbRC scores (1-2) in BV patients after treatment are indicators of recurrence, and whether preemptive action, based on this score, with more intensive treatment, delays or eliminates recurrence in these patients.

DETAILED DESCRIPTION:
A standard of care (SOC) treatment for BV is oral metronidazole 500 mg twice a day for 7 days (8). The investigators will use this for all enrollees with BV as the initial treatment. The investigators will evaluate patients at each visit by LbRC scores; a score of 1-2 (low) indicates that notable levels of non-lactobacilli are present. BV subjects with clinical cures (Amsel) and LbRC scores of 3-4 (high) at Visit 2 will simply be monitored on a monthly basis with no further treatment (Group G1). The investigators expect that some Group 1 patients will eventually recur, and that LbRC scores will drop to 1-2, two weeks prior to recurrence of BV symptoms, an event the investigators termed "conversion" . The investigators will choose randomly, using an Excel randomizer, half of the "converted" patients (Group G2) to be treated with a high dose metronidazole (HDM) regimen, one 750 mg metronidazole/ 200 mg miconazole vaginal suppository daily for 7 days, to determine if treatment initiated by the LbRC "warning" prevents recurrence. These randomized and re-treated Group G2 subjects will be moved to Group B2.

Patients who are "cured" by Amsel criteria and Nugent score but not by LbRC score at Visit 2, will be randomly divided into 2 groups per pre-randomization code the laboratory has. One (B1 Group) will be monitored monthly for up to 9 months for recurrence, with no further treatment in that interval. Another group (B2) will be randomized to receive the HDM treatment, and will be monitored for long term recurrence for up to 9 months. The Lab will notify the nurse as to which study number subject has been randomized to be retreated with HDM. The nurse will contact the subject to come in for a urine pregnancy test and for the medication and instructions on its use. All subjects will be asked to obtain daily vaginal samples, which will be stored at room temperature and returned at the next visit where more supplies will be obtained. Subjects will continue taking daily specimens for as long as the subject is enrolled and willing to do so. All subjects who return the daily samples will be compensated for their time with a $25 Target gift card at each visit.

Fifty non-BV subjects with no history of "vaginitis" in the past year will be enrolled as a control Group H and seen monthly to monitor the LbRC in the vaginal secretions. All subjects will be asked to take daily dated vaginal samples and store them in supplied containers at room temperature and return the vaginal swabs at each monthly visit where they will receive more supplies for the next month of specimens. All subjects will be compensated with a $25 gift card from Target at each scheduled visit for their time and the return of the vaginal swab samples.

Subjects in Group G1 or B1 who recur with acute symptomatic BV, and randomly half of those in Group G1 who "convert" from a good LbRC score to a poor LbRC score without symptoms, will be offered to take the 7 day HDM vaginal suppository regimen for one time only. Should the subject relapse after taking the HDM vaginal suppositories, she will be dropped from the study and given a prescription for conventional or SOC treatment of her BV. Should a subject return with a trichomonas infection she will be dropped from the study and treated with prescription medication. Should a subject return with vulvovaginal candidiasis, she will be given a prescription for an anti-yeast medication and may continue in the study.

Purpose of the study:

Diagnosis: Is the sensitivity, specificity, positive and negative predictive value of LbRC equal to or better than Nugent Score or commercial tests (BD Affirm VIII, BV Blue, targeted qPCR)? Prognosis and individualized therapy: Does a poor LbRC score in post-treatment, "cured" BV patients predict more rapid recurrence? Does intervention with more rigorous treatment, based on this score, delay or prevent recurrence? The proposed pilot study is a randomized pilot, prospective study that will will enroll at least 50 healthy women and 140 women with acute to recurrent BV

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria For BV Subjects: (140 subjects)

* Premenopausal women over the age of 18 who have BV who are willing to sign informed consent.
* Positive for all Amsel criteria:

  * Vaginal pH > 4.5
  * Positive amine test
  * > 20% clue cells on wet mount
  * Grayish-white adherent discharge
* Subject is willing to refrain from using any vaginal medications, douches or spermicides except for the metronidazole suppositories that are given to her for the duration of the study.
* Subject is willing to use supplied non-lubricated condoms when sexually active. But not to have sexual intercourse within 48 hours of any Study Visit.
* Subject to refrain from alcohol for 24 hours prior to the first 7 days of the metronidazole treatment and for 48 hours after completion of this treatment.

Inclusion criteria for Healthy control group.

* Enrollees for the healthy Group H in the study must be premenopausal and have not experienced any vaginitis in the past year.
* Subject will be encouraged to have a full clinical examination, but if she declines, she must have a self-swab evaluation that is normal (no yeast, no clue cells, normal flora, no parabasal cells and no trichomonads) and will be retained in Group H if her Nugent score is 3 or less.
* Subject must be willing to obtain daily samples and return monthly with the samples for a self-swab evaluation and a replenishment of the daily swab supplies. Healthy women will continue for as long as they are willing up to 9 months.
* Healthy women will be asked to use the supplied non-lubricated condoms, but will not be dropped from the study if they do not.
* Must be using some form of contraception if sexually active.

Exclusion Criteria:

Study Exclusion Criteria for BV Study Subjects:

* Mixed vaginal infection at time of enrollment.
* Pregnancy, nursing or planning on getting pregnant.
* Subject on anticoagulation therapy, lithium therapy or Antabuse therapy.
* Vaginal bleeding at time of enrollment
* Allergy to metronidazole
* Use of any vaginal antibiotics or antifungals in the previous 10 days, from enrollment.
* Must not require treatment for an abnormal Pap smear or genital cancer.
* Must abstain from vaginal douching during enrolled period.

Study Exclusion for Control Subjects:

* Has a vaginal infection at enrollment
* Pregnant, nursing or planning on becoming pregnant in the next year.
* Vaginal bleeding at enrollment
* Must not require treatment of any genital cancer or abnormal pap smear
* Should abstain from douching throughout the length of the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of bacterial vaginosis | Monthly for up to nine months
  Patients and control women will be assessed monthly for bacterial vaginosis by Nugent and Amsel criteria

SECONDARY OUTCOMES:
Relative quantity of Lactobacillus among total vaginal bacteria | Monthly clinical visits and daily swabs for up to nine months
  This quantitative assay of relative Lactobacillus content of vaginal swabs will be assessed monthly by qPCR, from samples taken at the clinic and from daily self swabs. This will be reported as a score, which is proportional to percentage Lactobacillus, and also integrates a score which reflects the prevalence of mid to low levels of non-Lactobacillus species.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Akins, PhD, Principal Investigator — Wayne State University; Jack D Sobel, MD, Principal Investigator — Wayne State University
Locations (1):
- WSU Tolan Park Medical Building 3901 Chrysler Service Drive, Suite 4A, Detroit, Michigan, United States

REFERENCES:
- [Background] Aguin T, Akins RA, Sobel JD. High-dose vaginal maintenance metronidazole for recurrent bacterial vaginosis: a pilot study. Sex Transm Dis. 2014 May;41(5):290-1. doi: 10.1097/OLQ.0000000000000123. PMID 24722380
- [Background] Aguin TJ, Akins RA, Sobel JD. High-dose vaginal metronidazole for recurrent bacterial vaginosis--a pilot study. J Low Genit Tract Dis. 2014 Apr;18(2):156-61. doi: 10.1097/LGT.0b013e31829a5558. PMID 23994951
- [Background] Lambert JA, John S, Sobel JD, Akins RA. Longitudinal analysis of vaginal microbiome dynamics in women with recurrent bacterial vaginosis: recognition of the conversion process. PLoS One. 2013 Dec 20;8(12):e82599. doi: 10.1371/journal.pone.0082599. eCollection 2013. PMID 24376552
- [Background] Lambert JA, Kalra A, Dodge CT, John S, Sobel JD, Akins RA. Novel PCR-based methods enhance characterization of vaginal microbiota in a bacterial vaginosis patient before and after treatment. Appl Environ Microbiol. 2013 Jul;79(13):4181-5. doi: 10.1128/AEM.01160-13. Epub 2013 Apr 26. PMID 23624483